CLINICAL TRIAL: NCT07094503
Title: Improving Access to Services, Preventing Eating Disorders, and Addressing Comorbid Depression and Anxiety in Diverse Adolescents
Brief Title: Adolescent Chatbot
Acronym: EMBody
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ellen E. Fitzsimmons-Craft, Associate Professor of Psychological & Brain Sciences, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202501059
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Body Image Disturbance; Disordered Eating Behaviors; Eating Disorder Prevention
Keywords: Adolescents; Disordered Eating Behaviors; Eating Disorder Symptoms; Eating Pathology; Eating disorder Prevention; Body Image; Body Image Disturbance; Digital Mental Health; Chatbot
MeSH Terms: conditions — Disordered Eating Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot Intervention Condition (Experimental): Participants receive access to the digital chatbot program featuring 5 CBT based modules for 3 months. Modules include psychoeducation and CBT-based exercises on regular eating and improving body image.
  Interventions: Behavioral: Wysa Digital Chatbot Program
- Waitlist Control (No Intervention): Participants receive access to the digital chatbot program after 6 months and completion of the study.

INTERVENTIONS:
Behavioral: Wysa Digital Chatbot Program — Wysa is a digital rules-based chatbot program platform offering cognitive-behavioral therapy-based guided self-help modules, including five modules for eating and body image developed by our team. Participants in this arm will engage with the digital chatbot program daily for three months to complete all five modules.
  Arms: Chatbot Intervention Condition

SUMMARY:
The purpose of this study is to test an eating disorders prevention digital chatbot program in a diverse group of adolescents.

DETAILED DESCRIPTION:
Eating disorders (EDs) are impacting youth at extreme rates, with up to 22% of adolescents reporting ED symptoms, and are associated with very high psychiatric comorbidity. Since adolescence is a critical period for the onset of eating disorders, prevention during this stage is essential to reducing lifetime prevalence. Interventions have been developed to prevent the onset of these devastating disorders, but these programs are generally not publicly available and rarely offer support for addressing comorbidity or the unique needs of vulnerable subpopulations (e.g., low-income populations, sexual and gender minorities, racial/ethnic minorities, those from rural areas), who are even less likely to have access to high-quality care. One scalable, engaging, easy-to use, and convenient approach to increasing access to evidence-based EDs prevention for underserved groups involves using a chatbot. This project will adapt our team's existing EDs prevention chatbot for use with adolescents, including those from diverse backgrounds, and evaluate its effectiveness. Our deep industry and non-profit partnerships will ensure scalability and ultimate real-world impact.

ELIGIBILITY:
Inclusion Criteria

1. 13 - 17 years old
2. Owns a smartphone
3. Speaks English
4. US resident
5. Screens as at-risk for an eating disorder
6. Not currently in treatment for an eating disorder

Exclusion Criteria:

1. Below 13 or older than 17 years of age
2. Does not own a smartphone
3. Does not speak English
4. Lives outside the US
5. Screens as:

   1. Having a subclinical or clinical ED
   2. Not at risk for an ED
   3. In treatment for an ED

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
ED risk factors; Weight Concerns Scale | 6 - months
  Weight concerns scale as found in the Stanford Washington Eating Disorder (SWED) screen is a 5-item validated self-report questionnaire which measures concern with weight and dieting. Each item is scored on a 5-100 scale, then an average is computed across all 5 items for a 0-100 score.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Fitzsimmons-Craft, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
The study is not federally funded.

REFERENCES:
- See also: Prescreen to the Study — https://washu.qualtrics.com/jfe/form/SV_0PX2BXw3bYrT1rM?Source=ClinTrials